CLINICAL TRIAL: NCT06647992
Title: Effect of Nurse Navigation Program on Cervical Cancer Screening Behaviour of the Women Aged 30-65
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TURKAN OZDAS (Other)
Responsible Party: Sponsor-Investigator, TURKAN OZDAS, Oncology Nursing PhD Student, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: SaglikBilimleriU-ON-TO-01
Record Dates: First submitted 2024-10-10; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancers
Keywords: Uterine Cervical Neoplasms; Patient Navigation; Transtheoretical Model; Health behavior
MeSH Terms: conditions — Uterine Cervical Neoplasms; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- Nurse Navigation Program (Experimental): The standard education and information booklet will be applied to both the experimental and control groups. Nurse navigation program will be applied to the experimental group. Within the navigation program, HPV DNA and Pap Smear Test Training and Counseling, Nurse Managed Telephone Support Line, Reminder Telephone Message, Transtheoretical Model and Motivational Interviews will be applied to individuals. Health Belief Model Scale for Cervical Cancer and Pap Smear Test: Psychometric testing is planned to be applied to both groups before and after the intervention in terms of outcome variables at 3 and 6 months.
  Interventions: Behavioral: Nurse Navigation Program
- control group- Standardised Education (No Intervention): It was planned to give "Cervical Cancer Education and Information Booklet" to the women in the control group about cervical cancer. Health Belief Model Scale for Cervical Cancer and Pap Smear Test: Psychometric testing was planned to be applied before and after the standard education and booklet in terms of outcome variables at 3 and 6 months.

INTERVENTIONS:
Behavioral: Nurse Navigation Program — It is planned to provide "Cervical Cancer Education and Counseling" to women in the experimental group about cervical cancer. Training and counseling is planned to be implemented face to face. An information booklet will be given to the experimental group. After 30 and 60 days after the training and counseling given to the experimental and control groups, it was planned to provide online (WhatApp) training and counseling to the patients in the experimental group:
  Participants will be given a contact number that they can reach during the day when they want to receive counseling about HPV-DNA or Pap smear. Interviews will be scheduled between 08.00-20.00.
  Individuals who are not screened will receive a reminder message by phone on the 45th and 75th day. Transtheoretical Model In the study, interventions will be planned for the experimental group according to the stages of the transtheoretical model.
  The researcher will conduct motivational interviews with the individuals.
  Arms: Intervention group- Nurse Navigation Program

SUMMARY:
This study was designed as a randomized controlled experimental study to examine the effect of the 'Nurse Navigation Program' on cervical cancer screening behaviors (Human Papilloma Virus (HPV) DNA screening test and/or pap smear test) and health beliefs about cervical cancer screening in women aged 30-65 years.

DETAILED DESCRIPTION:
An important step in the fight against cervical cancer is access to early diagnosis, early screening culture and the creation of screening opportunities. Problems in access to health services, barriers and cultural reasons play an important role in participation in cervical cancer screening. Nurse The Navigation Program is important to help individuals overcome and cope with these barriers. There are international studies showing the positive effect of the nurse navigation program on cervical cancer screening behaviors. However, it is thought that this study will contribute to the literature because the number of studies on this subject is not sufficient and no research is found in national sources.

It is aimed to contribute to overcoming the problems and obstacles in front of the patients' access to cervical cancer screening with the Nurse Navigation Program application developed based on the Transtheoretical Model to the experimental group and to provide evidence for the nurse navigation program application to be a method used in the cervical cancer screening process.

The population of the study will consist of female members of Non-Governmental Organizations in the 30-65 age group. The data of the study will be collected between September 13, 2024 and February 15, 2025 after ethics committee approval and institutional permission. The design of the study is a randomized controlled experimental study.

The data will be collected using the Individual Descriptive Information Form, Information Questions on Reproductive Health and Sexual Life, Questions on Cervical Cancer and Screening, Questions on HPV Knowledge, Cervical Cancer and Pap Smear Test Health Belief Model Scale. The statistical data obtained as a result of the research will be analyzed using the SPSS package program. It is expected that the rate of having HPV-DNA test and Pap smear test is higher in the experimental group in which the nurse navigation program is applied compared to the control group in which the intervention is not applied, and the mean score of benefit perception of cervical cancer screening behaviors (HPV DNA and/or Pap smear) is expected to be significantly different in the group in which the nurse navigation program is applied compared to the group in which it is not applied.

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years old,
* With health insurance,
* No history of gynecologic cancer,
* Current or past active sexual life
* Women who agreed to participate in the study

Exclusion Criteria:

* Diagnosed with gynecologic cancer,
* The one who had a hysterectomy,
* Who do not want to be involved in the study,
* No previous sexual experience,

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 80 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Health Belief Model Scale for Cervical Cancer and Pap Smear Test: Psychometric testing | Pre-test, 3rd month post-test, 6th month post-test
  Health Belief Model Scale for Cervical Cancer and Pap Smear Test: Psychometric testing consists of 35 items grouped into five subscales.
  1. Pap smear Benefit (items 18.-22.) and Health Motivation (items 11.-14.) subscales
  2. Pap smear Perception of obstacle (items 23-36) subscale,
  3. Cervical cancer severity perception (Items 4-10) subscale,
  4. Cervical cancer sensitivity perception (Items 1 - 3) subscale,
  5. Health Motivation subscale (items 15-17) A 5-point Likert scale ranging from 1 to 5 - "strongly disagree" (1), "disagree" (2), "undecided" (3), "agree" (4), "strongly agree" (5) - was used to assess the scale. Each dimension of the scale is evaluated separately and not combined into a single total score. For each individual, as many points are obtained as the number of sub-dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Turkan Ozdas, Principal Investigator — Saglık Bilimleri University; Donmez Elif, Study Director — Saglık Bilimleri University
Locations (1):
- Saglık Bilimleri University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No